CLINICAL TRIAL: NCT04744415
Title: Epidemiology of the Hospitalizations in the Italian Coronary Care Unit Network at the Time of Covid19
Brief Title: Hospitalizations During Pandemia in the Italian Coronary Care Unit Network
Acronym: BLITZ-COVID19
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K22
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Management and Epidemiology of Patients Admitted in ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Epidemiology of admissions — Cardiology Intensive Care Unit admission

SUMMARY:
Multicentre, national, observational, retrospective and prospective study.

The BLITZ-COVID19 study aims at describing the epidemiology of admissions to Italian Cardiology Intensive Care Units in the COVID-19 infection pandemia, the main aspects of the clinical management of inpatients, their short-term outcome, the absorption of resources related to their admission.

DETAILED DESCRIPTION:
The BLITZ-COVID19 study, aims at describing the epidemiology of admissions to Italian Cardiology Intensive Care Units .

The study is observational, multicentre, national and involves the collection of clinical data, both retrospectively and prospectively, using a web-based system. In conducting the study, no drugs are tested, nor are diagnostic tests or non-pharmacological therapies performed other than those that each participating cardiologist decides to perform following the rules of normal clinical practice. Diagnostic procedures and pharmacological and non-pharmacological therapies habitually prescribed for cardiovascular pathologies, which are the object of hospitalization, and those used in the event of a COVID-19 infection, will be recorded in the database.

ELIGIBILITY:
Inclusion Criteria:

- All patients aged ≥18 years admitted with any diagnosis to one of the participating ICU

Exclusion Criteria:

- Refuse to signe consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥18 years admitted with any diagnoses to ICU in the specified periods of 30 days each.
  Retrospecitve phase:(March 1-30, 2020 in the Northern or Centre-North regions; March 15-April 13, 2020 in the Southern or Ventre_South Regions and island.
  Perspective phase (depending by the IRB approval) in the following periods:
  November 9-December 8, 2020; November 23-December 22, 2020; January 11-February 9, 2021.
  (Retrospective study) or in the
Sampling Method: Probability Sample
Enrollment: 6054 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Impact that COVID-19 infection may have had on the in-hospital mortality | Enrollment
  Impact that COVID-19 infection may have had on the in-hospital mortality of the various clinical conditions admitted to ICU
Epidemiology and management of patients admitted to ICU | Enrollment
  The different diagnoses of discharge from the ICU and their frequency will be described. All hospitalized cardiac and non-cardiac pathologies will be listed, with particular reference to any COVID-19 infection.
Management of patients admitted to ICU | Enrollment
  Description of the main therapeutic decision in patients hospitalized for the most relevant pathologies

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Gulizia, MD, Study Chair — Heart Care Foundation
Locations (109):
- Italy (109):
  - Ospedale Santo Spirito - Sc Cardiologia, Casale Monferrato, AL
  - Istituto Scientifico Inrca - Uo Cardiologia/Utic/Telecardiologia, Ancona, AN
  - Ospedale Generale Regionale-Po U. Parini - U.O. Cardiologia E Cure Intensive Card., Aosta, AO
  - Po Sant'Ottone Frangipane - U.O.C. Cardiologia - Utic, Ariano Irpino, AV
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Ospedale Miulli - U.O.C. Cardiologia - Utic, Acquaviva delle Fonti, BA
  - Aou Policlinico - Uoc Cardiologia Ospedaliera, Bari, BA
  - Ospedale Di Venere - U.O.C. Di Cardiologia, Bari, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ospedale Di Bentivoglio - U.O. Di Cardiologia, Bentivoglio, BO
  - Ospedale Maggiore - U.O. Di Cardiologia, Bologna, BO
  - Asst Spedali Civili - Cardiologia, Brescia, BS
  - Ospedale Generale Regionale - Divisione Di Cardiologia, Bolzano, BZ
  - Arnas G. Brotzu - Cardiologia Con Utic, Cagliari, CA
  - A.O.U. Cagliari Policlinico Monserrato - Sc Cardiologia Utic Emodinamica, Monserrato, CA
  - Ospedale A. Cardarelli - U.O. Cardiologia E Utic, Campobasso, CB
  - Presidio Ospedaliero Moscati - U.O.C. Cardiologia-Utic, Aversa, CE
  - Az. Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia-Utic, Caserta, CE
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Presidio Ospedaliero San Rocco - U.O.C. Cardiologia - Utic, Sessa Aurunca, CE
  - Ospedale San Pio Da Pietrelcina - Cardiologia, Vasto, CH
  - Ospedale Regina Montis Regalis - U.O. Cardiologia-Utic, Mondovì, CN
  - Ospedale Maggiore Ss. Annunziata - Sc Cardiologia, Savigliano, CN
  - Ospedale Moriggia Pelascini - Unita' Operativa Di Cardiologia, Gravedona, CO
  - Ospedale S. Anna - U.O.C. Di Cardiologia, San Fermo della Battaglia, CO
  - P.O. Garibaldi Centro - U.O.C. Cardiologia, Catania, CT
  - Centro Cuore Morgagni - U.F. Utic Ed Emodinamica, Pedara, CT
  - Arcispedale Sant'Anna - U.O. Cardiologia - Utic, Ferrara, FE
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Ospedale Casa Sollievo Della Sofferenza - Cardiologia - Utic - Riabil Cardiologica, San Giovanni Rotondo, FG
  - Ospedale Santa Maria Annunziata - Cardiologia, Bagno a Ripoli, FI
  - Ospedale San Giuseppe - Cardiologia, Empoli, FI
  - Aou Careggi - Cardiologia Interventistica, Florence, FI
  - Ospedale San Giovanni Di Dio - Cardiologia, Florence, FI
  - Ospedale Santa Maria Nuova - Hdu Cardiologica/Utic, Florence, FI
  - E.O. Ospedali Galliera - S. C. Cardiologia, Genova, GE
  - Presidio Ospedaliero - U.O. Cardiologia, Sanremo, IM
  - Ospedale Civile Sacro Cuore Di Gesu' - Uo Cardiologia Utic, Gallipoli, LE
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic, Scorrano, LE
  - Azienda Osp. Cardinale G. Panico - U.O. Cardiologia - Utic, Tricase, LE
  - Ospedali Riuniti - U.O.C. Cardiologia E Utic, Livorno, LI
  - Nuovo Ospedale Versilia - Sc Cardiologia, Lido di Camaiore, LU
  - Ospedale San Gerardo - U.O. Cardiologia-Utic, Monza, MB
  - Aor Papardo - U.O. Cardiologia Con Utic, Messina, ME
  - Ospedale Piemonte - Cardiologia E Utic, Messina, ME
  - Centro Cardiologico Monzino - Terapia Intensiva Cardiologica (Utic), Milan, MI
  - Irccs Policlinico Multimedica - Uo Di Cardiologia, Sesto San Giovanni, MI
  - Ospedale Civile Di Baggiovara - U.O. Di Cardiologia, Modena, MO
  - Aou Maggiore Della Carita' - Cardiologia Ii, Novara, NOVARA
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Fondazione G. Giglio - U.O. Cardiologia E Utic, Cefalù, PA
  - Aor Villa Sofia-Cervello P.O. Cervello - U.O. Cardiologia - Cervello, Palermo, PA
  - Aor Villa Sofia-Cervello Po Villa Sofia - U.O.C. Cardiologia E Utic - Villa Sofia, Palermo, PA
  - Ospedale Civile 'Guglielmo Da Saliceto' - Uo Cardiologia, Piacenza, PC
  - Ospedale Civile Dello Spirito Santo - Utic E Cardiologia Interventistica, Pescara, PE
  - Presidio Ospedaliero Citta' Di Castello - U.O. Di Cardiologia, Città di Castello, PG
  - Ospedale Gubbio-Gualdo Tadino - U.O. Di Utic E Cardiologia, Gubbio, PG
  - Ospedale Generale Provinciale Lotti - U.O. Malattie Cardiovascolari Vde E Avc, Pontedera, PI
  - Ospedale Di Pordenone - S.O.C. Cardiologia, Pordenone, PN
  - Ospedale Santo Stefano - U.O. Cardiologia, Prato, PO
  - Ospedale Ss. Cosma E Damiano - U. O. Cardiologia - Utic, Pescia, PT
  - Ospedale Generale Di Zona - U.O. Cardiologia - Utic, Lagonegro, PZ
  - Azienda Ospedaliera San Carlo - Ssd Utic, Potenza, PZ
  - Ospedale Per Gli Infermi - U.O. Cardiologia - Utic, Faenza, RA
  - Ospedale Civile Santa Maria Delle Croci - U.O. Di Cardiologia, Ravenna, RA
  - P.O. San Camillo de Lellis - U.O.C. Cardiologia, Rieti, RI
  - Ospedale Civile San Paolo - U.O. Cardiologia - Utic, Civitavecchia, RM
  - Ospedale S. Maria Goretti - Uoc Malattie Cardiovascolari, Latina, RM
  - Aurelia Hospital - U.O.C Cardiologia, Roma, RM
  - Clinica Citta' Di Roma - Cardiologia-Utic, Roma, RM
  - European Hospital - U.O. Cardiologia Interventistica, Roma, RM
  - Ospedale Fatebenefratelli - U.O.C. Cardiologia, Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia, Roma, RM
  - Ospedale Sandro Pertini - Uoc Cardiologia, Roma, RM
  - Ospedale Sant'Andrea Di Roma - U.O.C. Cardiologia, Roma, RM
  - PO San Filippo neri - ASL Roma1, Roma, Roma
  - Ospedale Santa Maria Della Misericordia - U.O.C. Cardiologia, Rovigo, RO
  - Presidio Osped. S. Maria Della Speranza - U.O. Di Cardiologia, Battipaglia, SA
  - P.O. Nocera-Pagani - Osp. Umberto I - Uoc Cardiologia - Utic, Nocera Inferiore, SA
  - Presidio Ospedaliero Luigi Curto - Uo Cardiologia-Utic, Polla, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - U.O.C. Utic, Salerno, SA
  - Ospedale San Luca - U.O. Utic - Cardiologia, Vallo della Lucania, SA
  - Ospedale Dell'Alta Val D'Elsa - Uosd Cardiologia-Utic, Poggibonsi, SI
  - Aou Senese Ospedale S. Maria Alle Scotte - U.O.C. Cardiologia Clinico-Chirurg. Utic, Siena, SI
  - Ospedale Civile - U.O. Cardiologia, Sondrio, SO
  - Ospedale S. Andrea - S.C. Cardiologia, La Spezia, SP
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale G. Di Maria - Cardiologia Utic, Avola, SR
  - P.O. Lentini - U.O. Di Cardiologia Con Utic, Lentini, SR
  - Ospedale Nostra Signora Di Bonaria - U.O.C. Cardiologia E Utic, San Gavino Monreale, SU
  - Ospedale Santa Maria Del Carmine - Cardiologia, Rovereto, TN
  - Ospedale Santa Chiara - Divisione Di Cardiologia, Trento, TN
  - Po S. Antonio Abate Di Trapani - U.O.C. Di Cardiologia E Utic, Erice, TP
  - Ospedale Santa Maria Dei Battuti - U.O. Di Cardiologia, Conegliano, TV
  - Pou Santa Maria Della Misericordia - S.O.C. Cardiologia, Udine, UD
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Civile - U.O. Cardiologia, Mirano, VE
  - Ospedale Civile - U.O.C. Cardiologia, Arzignano, VI
  - Ospedale Civile San Bortolo - U.O.C. Cardiologia, Vicenza, VI
  - Casa Di Cura Dr. Pederzoli - Servizio Di Cardiologia, Peschiera del Garda, VR
  - Ospedale Ss. Trinita' - S.C. Di Cardiologia, Borgomanero
  - Ospedale San Leonardo - U.O. Di Cardiologia-Utic, Castellammare di Stabia
  - Ospedale San Giovanni Di Dio - Uo Cardiologia - Utic, Frattamaggiore
  - Ospedale Generale Di Zona - U.O. Cardiologia - Utic, Giugliano in Campania
  - Ospedale Anna Rizzoli - Cardiologia-Utic, Lacco Ameno
  - Aorn Cardarelli - U.O. Cardiologia Con Utic, Napoli
  - Clinica Mediterranea - U.O. Di Cardiologia, Napoli
  - Ospedale Del Mare - U.O. Cardiologia Con Utic, Napoli
  - Pres. Ospedaliero S. Maria Della Pieta' - U.O. Cardiologia E Utic, Nola

IPD SHARING:
Plan to Share IPD: Undecided
Still to be decided

REFERENCES:
- [Result] Gulizia MM, Fabbri G, Lucci D, Di Pasquale G, Gabrielli D, Campodonico J, Mauro A, Inciardi R, Di Lorenzo E, Oliva F, Nardi F, Colivicchi F, De Luca L; BLITZ-COVID19 Investigators. Type of hospitalisations and in-hospital outcomes in the Italian coronary care unit network at the time of COVID-19 pandemic: the BLITZ-COVID19 Registry. BMJ Open. 2022 Nov 29;12(11):e062382. doi: 10.1136/bmjopen-2022-062382. PMID 36446450